CLINICAL TRIAL: NCT04325464
Title: Open-label, 9-week Treatment, De-centralized Trial to Collect Real World Evidence for a Digital Therapeutic (DT) Delivering Cognitive Behavioral Therapy for Insomnia (CBT-I) for Participants With Chronic Insomnia
Brief Title: A Remote, 9-week Insomnia Treatment Trial to Collect Real World Data for a Digital Therapeutic
Acronym: DREAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pear Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEAR-003-101; DREAM Study (Other: Pear Therapeutics)
Record Dates: First submitted 2020-02-20; First posted 2020-03-27 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Chronic Insomnia
Keywords: Digital Therapeutic; CBT-I; Chronic Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- PEAR-003A (Experimental): Digital Therapeutic
  Interventions: Device: PEAR-003A

INTERVENTIONS:
Device: PEAR-003A — PEAR-003A delivers CBT-I through a decentralized clinical trial open to participants with chronic insomnia

SUMMARY:
The purpose of the study is to collect data in a real-world environment, for a digital therapeutic that delivers CBT-I through a decentralized clinical trial, open to participants with chronic insomnia.

DETAILED DESCRIPTION:
This is an open-access, open-label, decentralized clinical trial to collect real-world evidence for PEAR-003A, a digital therapeutic delivering CBT-I.

Potential participants will answer an online prescreening questionnaire to determine eligibility. Qualifying participants will proceed to complete 6 weekly modules through their personal mobile phone or tablet in nine weeks. A series of the assessment and questionnaires will be administered at set points during the study. Participants will be asked to complete a follow-up module about 26 weeks, and at Days 243 (6-month), 428 (12-month), 610 (18-month) and 793 (24-month) after completing treatment.

A subset of approximately 34 participants may be asked to partake in a optional user experience sub study. The participant will be asked to provide study feedback by either completing a five-day diary or an interview.

ELIGIBILITY:
Inclusion Criteria:

1. Provide electronic informed consent prior to any study specific assessments being performed
2. Between 22 and 75 years old, inclusively
3. Insomnia as defined by an ISI score of 8 or above
4. Insomnia symptoms for at least 3 months
5. < or = 6.5 hours of sleep per night
6. Access to a mobile device
7. Resident of the United States and currently living in the United States for the duration of the trial.

Exclusion Criteria:

1. Presence of an active and/or progressive physical illness (e.g., congestive-heart failure, chronic obstructive pulmonary disease, acute pain), neurological disorder (e.g., epilepsy) or neurological degenerative diseases (e.g., dementia, multiple sclerosis)
2. Unstable medication regimen (change to schedule or dosage within the past 3 months)
3. Diagnosis of a psychotic disorder or bipolar disorder or medical condition contraindicated by sleep restriction
4. Have family or work schedules that prevent them from having normal sleep schedules defined as bedtime between 8:00 pm and 2:00 am and/or waking times between 4:00 am and 10:00 am.
5. Individuals who need to be alert or cautious to avoid serious accidents in their job or daily life. Examples include: Long-haul truck drivers, Long-distance bus drivers, Air traffic controllers, Operators of heavy machinery, some assembly line jobs.
6. Pregnant or planning to become pregnant during the course of the trial.
7. Other untreated sleep disorders as self-reported by the participant (e.g., obstructive sleep apnea, periodic leg movements, parasomnias)
8. Participated in an investigational research study in the past 30 days

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1590 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index (ISI) | From Baseline to Day 63 (End of Treatment) and Days 243, 428, 610, 793 (Follow-up)
  Change in the Insomnia Severity Index's (ISI) total score from Baseline to End of Treatment and Follow-up. The ISI's total score ranges from 0 (not clinically significant) to 28 (clinically significant)

SECONDARY OUTCOMES:
Evaluate PEAR-003A Engagement Data | Baseline, Day 63, Day 243, Day 428, Day 610, Day 793
  Evaluate PEAR-003A engagement rates
Evaluate PEAR-003A Adherence Data | Baseline, Day 63, Day 243, Day 428, Day 610, Day 793
  Evaluate PEAR-003A adherence rates
Examine change in depression symptoms | Baseline, Day 63, Day 243, Day 428, Day 610, Day 793
  Change in the eight-item Patient Health Questionnaire (PHQ-8) scores from Baseline to End of Treatment and Follow-up. The PHQ's total score ranges from 0 (not clinically significant) to 24 (clinically significant)
Examine change in anxiety symptoms | Baseline, Day 63, Day 243, Day 428, Day 610, Day 793
  Change in the Generalized Anxiety Disorder-7's (GAD-7) scores from Baseline to End of Treatment and Follow-up. The GAD-7's total score ranges from 0 (not clinically significant) to 21 (clinically significant)

OTHER OUTCOMES:
Examine treatment responders' data | Baseline, Day 63, Day 243, Day 428, Day 610, Day 793
  Treatment responders are those whose ISI decreased by more than 7 points. Responders ISI score will be evaluated at the end of treatment and follow-up.
Examine Insomnia Remission | Day 63, Day 243, Day 428, Day 610, Day 793
  Subjects in treatment remission are those whose ISI score is 8 or less. Subjects in treatment remission ISI scores will be evaluated at end of treatment and follow-up
Describe user experience surveys | Baseline, Day 63
  Summarize user experience surveys through descriptive statistics
Describe user experience diary data | Baseline, Day 63
  Summarize qualitative diary data through descriptive statistics
Describe user experience interviews | Baseline, Day 63
  Summarize user experience interviews through descriptive statistics
To determine if there is a change in daytime sleepiness | Baseline, Day 63, Day 243, Day 428, Day 610, Day 793
  Change in Epworth Sleepiness Scale from baseline to end of treatment and follow-up. The ESS total score ranges from 0 (not clinically significant) to 24 (clinically significant)
To determine change in quality of life | Baseline, Day 63, Day 243, Day 428, Day 610, Day 793
  Change in quality of life as measured in The Short Form 12 (SF-12). The SF-12 summary scores range from 0-100 with higher scores representing better self-reported health
To determine change in work attendance and productivity | Baseline, Day 63, Day 243, Day 428, Day 610, Day 793
  Change in presenteeism/absenteeism work questions based on a survey. Subject answers Yes/No questions of whether continuously employed during the time period. If not, they can enter number of days employed or missed. Survey also contains a question regarding rating of productivity in %.
To evaluate potential changes in healthcare utilization and costs identified in claims | Matched period
  Change in tokenized health claims from a specified period (up to 24 months) prior to intervention and a similar period after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Abby Doctolero, Study Director — Pear Therapeutics, Inc.
Locations (1):
- Pear Therapeutics, Inc., Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thorndike FP, Morin CM, Ojile J, Edington S, Gerwien R, Ong JC, Wickwire EM, Ritterband LM, Riney H. Effect of a prescription digital therapeutic for chronic insomnia on post-treatment insomnia severity, depression, and anxiety symptoms: results from the real-world DREAM study. Front Psychiatry. 2024 Sep 10;15:1450615. doi: 10.3389/fpsyt.2024.1450615. eCollection 2024. PMID 39319356
- [Derived] Thorndike FP, Berry RB, Gerwien R, Braun S, Maricich YA. Protocol for Digital Real-world Evidence trial for Adults with insomnia treated via Mobile (DREAM): an open-label trial of a prescription digital therapeutic for treating patients with chronic insomnia. J Comp Eff Res. 2021 May;10(7):569-581. doi: 10.2217/cer-2021-0004. Epub 2021 Mar 8. PMID 33682430